CLINICAL TRIAL: NCT05254301
Title: Faster Functional Performance Recovery After Individualized Nutrition Therapy Combined With a Patient-tailored Physical Rehabilitation Program Versus Standard Physiotherapy in Patients With Long COVID: a Pilot Study.
Brief Title: Nutrition and LOComotoric Rehabilitation in Long COVID-19
Acronym: UNLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Waele, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-EDW-01; LCOV21-1306 (Other Grant/Funding Number: KCE)
Record Dates: First submitted 2022-02-19; First posted 2022-02-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: Nutrition; Pilot Study; Physical Therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized multimodal treatment (Experimental): A combination of biometric parameter oriented nutritional counseling and a tailored physical training program.
  Interventions: Other: Intervention group
- Standard care (Active Comparator): Physiotherapy with standard care advice for gradual cardiorespiratory and resistance training. (In this standard care setting, nutritional screening nor counseling is included.)
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — This personalised multimodal treatment considers evidence- and practice-based elements (e.g., self-management, individual guidance & follow-up, low-threshold activities, homebased functional training & better follow-up guidance afterwards).

SUMMARY:
Long COVID is a new phenomenon, in which individuals who experienced a SARS-CoV-2 infection still experience one or more symptoms, such as exercise intolerance, fatigue and/or muscle pains in addition to other COVID-related symptoms, weeks to months after initial infection.

The aim of this pilot-study is to learn about which complaints patients continue to experience after their infection and how this affects their lives to a greater or lesser extent and whether a patient-tailored physical rehabilitation programme combined with individualised nutritional therapy leads to a faster recovery compared to a classic exercise program with the physiotherapist.

DETAILED DESCRIPTION:
The rapid spread of SARS-CoV-2 virus has already led to more than 212 million confirmed cases. The acute phase of infection resulted in variable clinical presentations, from asymptomatic to severe illness requiring admission at an intensive care unit. As the COVID-19 pandemic evolves, long-term symptoms and functional problems related to the SARS-CoV-2 infection reached the surface. Approximately 5-10% of the infected people experience prolonged symptoms with predominant symptoms being overall reduced physical capacity, fatigue and muscle weakness. Exertional intolerance/post-exertional malaise is also frequently seen.

A growing group of patients experience persisting symptoms after the initial infection and these can have significant impact on daily functioning and quality of life. These patients feel 'abandoned' by healthcare providers and receive limited or conflicting advice. Treatment modalities for patients with long COVID have up and till now been scarcely investigated because there is insufficient understanding of the underlying mechanisms. However, most patients seek care and the majority of them receive physiotherapy/rehabilitation in one form or another in the 3 to 6 months after onset. Unfortunately, this seems not to be enough, on the contrary, patients seem to experience even more difficulties. Nutrition-wise, after highly prevalent weight loss in the active phase of COVID-19, challenges remain to improve protein intake and gain muscle mass. This stresses the need for a multidisciplinary approach and social support.

The aim of the current study is to investigate if a patient-tailored physical rehabilitation programme combined with nutritional optimisation with individualised therapy and counselling may lead to a faster improvement of functional performance compared to a standard physiotherapy programme in patients suffering from long-term effects (> 12 weeks) of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign written consent in Dutch, French or English
* Laboratory (PCR and/or serology) confirmed infection with SARS-CoV-2 less than 12 months ago
* Persisting functional difficulties and symptoms: exercise intolerance and/or fatigue and/or muscle pain beyond 12 weeks beside other COVID-related symptoms (e.g., loss of taste and/or smell)
* Patient affiliated to a social security system

Exclusion Criteria:

* Patients unable to comprehend oral and/or written instructions, questionnaires in English, French or Dutch.
* Patient currently suffers from any other disease beside long COVID that could explain the symptoms (e.g., fibromyalgia, Sjögren disease, severe anaemia...)
* Patient is unable to undergo a rehabilitation programme due to comorbidities (e.g., major cardiovascular disease such as myocarditis or severe dementia), as decided on by the medical study team members.
* Patient currently benefiting from physiotherapy sessions with focus on motor and/or respiratory therapy for COVID-19 or any other unrelated disease
* Patients with metabolic disorders or severe gastro-intestinal conditions (e.g. short bowel syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-04-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
1-minute sit-to-stand (1-MSTS) | Change from Baseline Repetitions Sit-To-Stand's in one minute at 12 weeks
  Testing of endurance and muscle strength of the lower extremities (standing up from a sitting position for as many repetitions as possible during 1 minute)

SECONDARY OUTCOMES:
Multi-dimensional Fatigue Inventor (MFI-20) | Change from Baseline MFI-20 at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  The MFI is a self-report instrument designed to measure fatigue and was initially developed in Dutch17 for patients with cancer. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue. It consists of 20 items divided over 5 dimensions (each 4 items) and is scored on a 5-point Likert scale. The higher the score the more severe the fatigue and by consequence the more impact fatigue has on daily functioning.
EuroQol five-dimensional (five-level version) (EQ-5D-5L) | Change from Baseline EQ-5D-5L at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Health-related Quality of Life will be measured by the EQ-5D-5L. This questionnaire comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels from no problems tot extreme problems. Next it contains a self-rated health status on a vertical visual analogue scale where the endpoints are labelled the best health you can imagine' and 'the worst health you can imagine'. This test has proven valuable for assessing physical health-related QoL (25).
Post-COVID-19 Functional Status (PCFS) | Change from Baseline PCFS at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Functional status will be evaluated for changes using the PCFS, specifically developed for COVID patients by Klok and colleagues.
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline HADS at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Mental status will be evaluated for differences using HADS.This test is a simple tool to assess both anxiety and depression, each with 7 questions.
Work Productivity and Activity Impairment (WPAI) | Change from Baseline WPAI at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Work capability will also be assessed using the Work Productivity and Activity Impairment. With 6 questions it asks about the decline in productivity and activity in the past 7 days. There are 3 versions available but all evaluate on absence, presence, loss of productivity and decline of activities during work. The WPAI is considered the best validated questionnaire for determining health-related work productivity and has been validated in various chronic inflammatory diseases.

OTHER OUTCOMES:
Muscle strength | Change from Baseline muscle strength at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Measurement of muscle strength by a handheld dynamometer (MicroFet).
Handgrip strength | Change from Baseline handgrip strength at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Measurement of handgrip strength using a JAMAR Hand Dynamometer
6-minute walk test (6-MWT) | Change from Baseline 6-MWT at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Testing functional status and fitness, and endurance (walking as far as possible for 6 minutes measuring total distance (meters)).
modified Medial Research Council (mMRC) | Change from Baseline mMRC at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Dyspnoea will be evaluated by the modified Medical Research Council.The participants answer the question if they sometimes feel short of breath. If so, they choose the quote that fits them most (score 0 "I feel only short of breath when performing heavy activities" to 4 "I am too short of breath to leave the house or I feel wheezy during dressing and undressing").
Barthel Index | Change from Baseline Barthel Index at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  The Barthel Index assesses to which extend a person needs help performing activities of daily living (ADL). Classical it consists of 10 items (but other versions exist) each scored for 0 to 1,2,3 on a total of 20. The higher the score the less dependent the individual.
Adequacy of feeding | Change from Baseline Adequacy of feeding at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Adequacy of feeding is the ratio between intake of calories and proteins and the individual need. The amount of proteins, carbohydrates and fatty acids to be eaten by the patient to fulfill the needs, are calculated based on the measured body weight. The caloric target is defined by a metabolic measurement: indirect calorimetry. People can be defined as hypo-, normo- or hypermetabolic when the measured value is compared to a calculated predictive value (e.g. 25 kcal/kg body weight/day). In case that the indirect calorimetry cannot be performed (e.g., claustrophobia), the caloric target will be defined using the best fitting formula (e.g. WHO equations for BMI < 18.5 kg/m², Harris-Benedict equation for normal- and overweight patients). The daily intake is compared to these needs: feeding adequacy.
Phase angle | Change from Baseline phase angle at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  This parameter is measured by Bio Impedance Analysis (BIA). The phase angle is a measure of cell and thereby body vitality.
Fat-to-fat free mass ratio | Change from Baseline fat-to-fat free mass ratio at 12 weeks, at 6 weeks intervention, at 12 weeks, and at 6 weeks post-intervention.
  Fat-to-fat free mass ratio us an important characteristic of a human being as it compares fat mass to fat free mass which includes bone muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair ziekenhuis Brussel, Brussels, Belgium

REFERENCES:
- [Derived] Roggeman S, Jimenez Garcia BG, Leemans L, Demol J, Geers J, De Smedt A, Putman K, Schiltz M, Beckwee D, De Waele E. Functional performance recovery after individualized nutrition therapy combined with a patient-tailored physical rehabilitation program versus standard physiotherapy in patients with long COVID: a pilot study. Pilot Feasibility Stud. 2023 Sep 28;9(1):166. doi: 10.1186/s40814-023-01392-1. PMID 37759324